CLINICAL TRIAL: NCT04317547
Title: A Hybrid Effectiveness-Implementation Trial to Improve Safe Driving Among Teen Drivers With Traffic Violations
Brief Title: Translation Study of a Safe Teen Driving Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ginger Yang (Other)
Collaborators: University of Iowa (Other)
Responsible Party: Sponsor-Investigator, Ginger Yang, Principal Investigator, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 3
Record Dates: First submitted 2020-03-04; First posted 2020-03-23 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Drive; Adolescent Behavior; Risk Behavior
MeSH Terms: conditions — Adolescent Behavior; Risk-Taking

STUDY DESIGN:
Intervention Model Description: We propose a hybrid, RCT to test the effectiveness and implementation of an evidence-based, parent-focused intervention among teen drivers with a moving violation. We aim to recruit 90 dyads (45 per group, totaling 180 study participants), comprised of one teen driver ages 16 or 17 who has committed a moving violation (e.g., speeding, failure to obey traffic signal) and the parent/legal guardian ('parent') who is most involved with the teen's driving. Recruitment will occur at the Franklin County Juvenile Traffic Court in Ohio following the parent-teen dyad's mandatory court appearance. After completing informed consent/assent and the baseline assessment, enrolled parent-teen dyads will be randomly assigned into either the Control or Intervention Group using a stratified block randomization. All enrolled dyads will be followed for a 6-month period.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): The Azūga™ in-vehicle driving feedback technology will be installed.32 This driving feedback technology consists of a pager-sized device plugged into the vehicle's on-board diagnostic (OBD) port (installed in the teen's car) and a smartphone app (downloaded on the teen's smartphone). All feedback features will be disabled. Control dyads will receive no driving feedback. The parent will not receive STS. Additionally, a wireless mini-camera will be installed on the dashboard in teen's car to identify the participating driver using facial verification technology.
- Intervention Group (Experimental): Parents will receive STS, which will include 1) Individualized virtual communication training and a booster session delivered by a traffic safety communication specialist; and 2) An online parent-teen safe driving communication guide. In addition, the Azūga™ in-vehicle device and app will be installed as described above and all feedback features will be enabled. Three types of feedback will be provided to teens: 1) Direct audio feedback; 2) Detailed cumulative driving data; and 3) A customized weekly driving summary report. Parents in this group will receive access to the teen's cumulative driving data and a weekly driving summary report. Additionally, a wireless mini-camera will be installed on the dashboard in teen's car to identify the participating driver using facial verification technology.
  Interventions: Behavioral: Steering Teens Safe (STS); Behavioral: Driving Feedback Technology.

INTERVENTIONS:
Behavioral: Steering Teens Safe (STS) — The goal of STS is to provide intervention parents with guidance and communication skills, which will enable parents to effectively communicate with their teens about specific driving safety topics (e.g., speeding, seatbelt use, distracted driving). Our proposed parent training has two components: an individualized virtual communication training (provided to parents via Skype by a trained research team member) and a parent-teen safe driving communication guide (available online).
  Other Names: STS
  Arms: Intervention Group
Behavioral: Driving Feedback Technology. — The driving feedback technology will include the Azūga™ in-vehicle device and smartphone app.
  Other Names: Azuga device
  Arms: Intervention Group

SUMMARY:
Steering Teens Safe (STS) is an evidence-based and parent-focused intervention developed by the investigators, which aims to improve safe teen driving practices by enhancing parental communication skills. The objective of this translation study is to assess the effect of STS on driving outcomes among teen drivers who have committed a traffic violation, and to assess the adoption and implementation fidelity of STS in a county court setting and among these high-risk teen drivers and their parents. The investigators will test the following specific aims: Aim 1: Determine the effects of the intervention on parent-teen communications and risky driving outcomes (risky driving events, unsafe driving behaviors, and recidivism) among teen drivers with a traffic violation(s). Aim 2: Assess the adoption of the intervention and implementation fidelity We will enroll 90 parent-teen dyads, comprised a teen driver (16 to 17 years) who committed a moving violation and a parent/legal guardian, from the Ohio Franklin County Juvenile Traffic Court following the teens' mandatory court hearing. Enrolled dyads will be randomly assigned to 1 of 2 study groups (n=45/group): 1) Control, device installation only with no feedback to nor communication training for parents, or 2) Intervention, device feedback to teens and parents, and parents will also receive individualized virtual communication training. The expected outcome is to establish the effectiveness of STS augmented with driving feedback technology, and to establish the implementation fidelity of STS in a court setting.

DETAILED DESCRIPTION:
Motor vehicle collisions (MVCs) are the leading cause of death among teenagers in the United States. Teen drivers who have committed a traffic violation are at an even greater risk for MVCs than their counterparts. While parent-focused interventions are an effective strategy to improve teen driving safety, most of these interventions target teen drivers are implemented as universal interventions (for teens of all risk profiles). Evidence on the effectiveness of these evidence-based interventions when translated and implemented among high-risk teen drivers such as those with a traffic citation is lacking.

The current project is significant because it will translate the STS program to the needs of high-risk teen drivers who have committed a traffic violation and their parents. This study is innovative because it partners with the local court system, and utilizes novel and cutting-edge in-vehicle technology. The findings of the current study will have a significant impact on juvenile traffic court's practices and policies aimed to improve teen driving safety by reducing MVC-related crashes, injuries, and deaths.

ELIGIBILITY:
Inclusion Criteria:

* Age 16-17 years at time of violation;
* Convicted of a moving violation;
* Possess a valid intermediate driver's license issued by the state of Ohio, with proof of car insurance;
* Access to a vehicle with an On-board Diagnostics II system port (i.e., cars made after 1996) in which he/she is the primary driver;
* Smartphone with Bluetooth capabilities;
* At least one legal guardian.

Exclusion Criteria:

* Unable to drive due to injury, license suspension, or car damage;
* Vehicle already has an in-vehicle driving feedback system installed;
* Extremely low average weekly drive time (e.g. <1 hour per week);
* Currently enrolled in another driving-related study;
* Ward of the State;
* Non-English speaking parent.

Ages: 16 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 180 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Frequency of Parent-teen communications | Six months/study period
  Frequency of parent-teen communication about driving safety. This will be measured through a survey asking parents how often they discussed the topic with their teen on driving topics.
Number of Risky driving events and unsafe behavior rates | Six months/study period
  Events of hard braking, sudden acceleration, speeding, distracted driving, and no seatbelt use.
Recidivism | Up to one year post-study period
  Recidivism will be measured among teens in both groups by linking traffic citations and court disposition data with the participating teen's driver's license number. Recidivism during the 12 months following enrollment, including date and type of violation, and days from index violation to subsequent violation will be analyzed
Adoption of the intervention | Six months/study period
  Adoption of the intervention by using publicly available court data from Franklin County Juvenile Traffic Court and compare it to all other juvenile traffic courts in Ohio. We will also use participant characteristic data and compare it to non-participating teens with a moving violation in Ohio.
Implementation fidelity | Six months/study period
  Engagement with community training via a self-report questionnaire, engagement with device feedback via Google Analytics, and a fidelity checklist will be combined to report implementation fidelity
Quality of Parent-teen communication | Six months/study period
  The quality of parent-teen communication about driving safety will be measured through an average rating of each driving topic which is recorded by the parent and teen.

CONTACTS AND LOCATIONS:
Overall Officials: Jingzhen (Ginger) Yang, PhD, MPH, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data used and/or analyzed during the current study, along with detailed study protocol, are available from the PI, Dr. Jingzhen Yang, on reasonable request. The data are not publicly available due to privacy restrictions.
Supporting Information: Study Protocol, SAP
Time Frame: Starting 6 months after the summary data are published.
Access Criteria: De-identified data collected for the study and a data dictionary will be made available to other researchers following approval of a study proposal by the PI, Dr. Jingzhen Yang (ginger.yang@nationwidechildrens.org) The study protocol, and statistical analysis plan are also available from the PI, Dr. Jingzhen Yang.

REFERENCES:
- [Background] Masten SV, Foss RD, Marshall SW. Graduated driver licensing and fatal crashes involving 16- to 19-year-old drivers. JAMA. 2011 Sep 14;306(10):1098-103. doi: 10.1001/jama.2011.1277. PMID 21917580
- [Background] Simons-Morton BG, Ouimet MC, Zhang Z, Klauer SE, Lee SE, Wang J, Albert PS, Dingus TA. Crash and risky driving involvement among novice adolescent drivers and their parents. Am J Public Health. 2011 Dec;101(12):2362-7. doi: 10.2105/AJPH.2011.300248. Epub 2011 Oct 20. PMID 22021319
- [Background] Mayhew DR, Simpson HM, Pak A. Changes in collision rates among novice drivers during the first months of driving. Accid Anal Prev. 2003 Sep;35(5):683-91. doi: 10.1016/s0001-4575(02)00047-7. PMID 12850069
- [Background] McCartt AT, Shabanova VI, Leaf WA. Driving experience, crashes and traffic citations of teenage beginning drivers. Accid Anal Prev. 2003 May;35(3):311-20. doi: 10.1016/s0001-4575(02)00006-4. PMID 12643948
- [Background] Insurance Institute for Highway Safety (IIHS). Fatality Facts: Teenagers 2015. Arlington (VA): The Institute; 2017 [cited 2018 Jan 4]. http://www.iihs.org/iihs/topics/t/teenagers/fatalityfacts/teenagers
- [Background] Rajalin S. The connection between risky driving and involvement in fatal accidents. Accid Anal Prev. 1994 Oct;26(5):555-62. doi: 10.1016/0001-4575(94)90017-5. PMID 7999200
- [Background] Summala H, Rajalin S, Radun I. Risky driving and recorded driving offences: a 24-year follow-up study. Accid Anal Prev. 2014 Dec;73:27-33. doi: 10.1016/j.aap.2014.08.008. Epub 2014 Aug 27. PMID 25171522
- [Background] Alver Y, Demirel MC, Mutlu MM. Interaction between socio-demographic characteristics: traffic rule violations and traffic crash history for young drivers. Accid Anal Prev. 2014 Nov;72:95-104. doi: 10.1016/j.aap.2014.06.015. Epub 2014 Jul 12. PMID 25019690
- [Background] Ayuso M, Guillen M, Alcaniz M. The impact of traffic violations on the estimated cost of traffic accidents with victims. Accid Anal Prev. 2010 Mar;42(2):709-17. doi: 10.1016/j.aap.2009.10.020. Epub 2009 Nov 22. PMID 20159098
- [Background] Factor R. The effect of traffic tickets on road traffic crashes. Accid Anal Prev. 2014 Mar;64:86-91. doi: 10.1016/j.aap.2013.11.010. Epub 2013 Dec 2. PMID 24342150
- [Background] Gebers MA, Peck RC. Using traffic conviction correlates to identify high accident-risk drivers. Accid Anal Prev. 2003 Nov;35(6):903-12. doi: 10.1016/s0001-4575(02)00098-2. PMID 12971925
- [Background] Goldenbeld C, Reurings M, Van Norden Y, Stipdonk H. Crash involvement of motor vehicles in relationship to the number and severity of traffic offenses. An exploratory analysis of Dutch traffic offenses and crash data. Traffic Inj Prev. 2013;14(6):584-91. doi: 10.1080/15389588.2012.743125. PMID 23859422
- [Background] Curry AE, Peek-Asa C, Hamann CJ, Mirman JH. Effectiveness of Parent-Focused Interventions to Increase Teen Driver Safety: A Critical Review. J Adolesc Health. 2015 Jul;57(1 Suppl):S6-14. doi: 10.1016/j.jadohealth.2015.01.003. PMID 26112737
- [Background] Beck KH, Shattuck T, Raleigh R. Parental predictors of teen driving risk. Am J Health Behav. 2001 Jan-Feb;25(1):10-20. doi: 10.5993/ajhb.25.1.2. PMID 11289724
- [Background] Hartos J, Eitel P, Simons-Morton B. Parenting practices and adolescent risky driving: a three-month prospective study. Health Educ Behav. 2002 Apr;29(2):194-206. doi: 10.1177/109019810202900205. PMID 11942714
- [Background] Simons-Morton B. Parent involvement in novice teen driving: rationale, evidence of effects, and potential for enhancing graduated driver licensing effectiveness. J Safety Res. 2007;38(2):193-202. doi: 10.1016/j.jsr.2007.02.007. Epub 2007 Mar 26. PMID 17478190
- [Background] Simons-Morton BG, Ouimet MC, Catalano RF. Parenting and the young driver problem. Am J Prev Med. 2008 Sep;35(3 Suppl):S294-303. doi: 10.1016/j.amepre.2008.06.018. PMID 18702985
- [Background] Zakrajsek JS, Shope JT, Greenspan AI, Wang J, Bingham CR, Simons-Morton BG. Effectiveness of a brief parent-directed teen driver safety intervention (Checkpoints) delivered by driver education instructors. J Adolesc Health. 2013 Jul;53(1):27-33. doi: 10.1016/j.jadohealth.2012.12.010. Epub 2013 Mar 6. PMID 23481298
- [Background] Goodwin AH, Foss RD, Margolis LH, Harrell S. Parent comments and instruction during the first four months of supervised driving: an opportunity missed? Accid Anal Prev. 2014 Aug;69:15-22. doi: 10.1016/j.aap.2014.02.015. Epub 2014 Mar 2. PMID 24641793
- [Background] Mirman JH, Albert WD, Curry AE, Winston FK, Fisher Thiel MC, Durbin DR. TeenDrivingPlan effectiveness: the effect of quantity and diversity of supervised practice on teens' driving performance. J Adolesc Health. 2014 Nov;55(5):620-6. doi: 10.1016/j.jadohealth.2014.04.010. Epub 2014 Jun 9. PMID 24925492
- [Background] Mirman JH, Curry AE, Winston FK, Wang W, Elliott MR, Schultheis MT, Fisher Thiel MC, Durbin DR. Effect of the teen driving plan on the driving performance of teenagers before licensure: a randomized clinical trial. JAMA Pediatr. 2014 Aug;168(8):764-71. doi: 10.1001/jamapediatrics.2014.252. PMID 24957844
- [Background] Simons-Morton BG, Hartos JL, Leaf WA, Preusser DF. Persistence of effects of the Checkpoints program on parental restrictions of teen driving privileges. Am J Public Health. 2005 Mar;95(3):447-52. doi: 10.2105/AJPH.2003.023127. PMID 15727975
- [Background] Ramirez M, Yang J, Young T, Roth L, Garinger A, Snetselaar L, Peek-Asa C. Implementation evaluation of steering teens safe: engaging parents to deliver a new parent-based teen driving intervention to their teens. Health Educ Behav. 2013 Aug;40(4):426-34. doi: 10.1177/1090198112459517. Epub 2012 Oct 4. PMID 23041706
- [Background] Peek-Asa C, Cavanaugh JE, Yang J, Chande V, Young T, Ramirez M. Steering teens safe: a randomized trial of a parent-based intervention to improve safe teen driving. BMC Public Health. 2014 Jul 31;14:777. doi: 10.1186/1471-2458-14-777. PMID 25082132
- [Background] Yang J, Campo S, Ramirez M, Krapfl JR, Cheng G, Peek-Asa C. Family communication patterns and teen drivers' attitudes toward driving safety. J Pediatr Health Care. 2013 Sep-Oct;27(5):334-41. doi: 10.1016/j.pedhc.2012.01.002. Epub 2012 Feb 22. PMID 22361241
- [Background] Winston FK, Mirman JH, Curry AE, Pfeiffer MR, Elliott MR, Durbin DR. Engagement with the TeenDrivingPlan and diversity of teens' supervised practice driving: lessons for internet-based learner driver interventions. Inj Prev. 2015 Feb;21(1):4-9. doi: 10.1136/injuryprev-2014-041212. Epub 2014 Jun 10. PMID 24916684
- [Background] McCartt AT, Farmer CM, Jenness JW. Perceptions and experiences of participants in a study of in-vehicle monitoring of teenage drivers. Traffic Inj Prev. 2010 Aug;11(4):361-70. doi: 10.1080/15389588.2010.486428. PMID 20730683
- [Background] Winston FK, Puzino K, Romer D. Precision prevention: time to move beyond universal interventions. Inj Prev. 2016 Apr;22(2):87-91. doi: 10.1136/injuryprev-2015-041691. Epub 2015 Aug 13. No abstract available. PMID 26271260
- [Background] Gielen AC, Frattaroli S, Pollack KM, Peek-Asa C, Yang JG. How the science of injury prevention contributes to advancing home fire safety in the USA: successes and opportunities. Inj Prev. 2018 Jun;24(Suppl 1):i7-i13. doi: 10.1136/injuryprev-2017-042356. Epub 2018 Feb 26. PMID 29483239
- [Background] Franklin County Court of Common Pleas. Meet the Magistrate. [Accessed 2018 Jan 4]. https://drj.fccourts.org/DRJ.aspx?PN=Susan_House.htm
- [Background] Peek-Asa C, Reyes M, Hamman C, Butcher B, Cavanaugh J. In-vehicle video feedback systems and parent engagement: a randomized trial to improve safe teen driving. Transportation Research Board. January 2016. Washington D.C.